CLINICAL TRIAL: NCT06757218
Title: Comparison of Autogenous Dentin Graft With Albumin Platelet Rich Fibrin Versus Autogenous Dentin Graft With Platelet Rich Fibrin in Alveolar Socket Preservation: A Randomized Controlled Clinical Trial.
Brief Title: Post Extraction Changes After Alveolar Socket Preservation Using Autogenous Dentin Graft (ADG) Combined With Either Albumin Platelet-rich Fibrin (ALB-PRF) or Standard Platelet-rich Fibrin (PRF).
Acronym: Alb-PRF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, MUATH ATIF MOHAMEDAHMED HASSAN, Master student, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-471
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Alveolar Socket Preservation
Keywords: Autogenous Dentin Graft; Albumin Platelet Rich Fibrin; Platelet Rich Fibrin

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical study, Double blinded (patients and biostatistician) with allocation ratio 1:1:1 using 3 - arm parallel groups (2 experimental and control).
Who Masked: Outcomes Assessor
Masking Description: Blinding is achievable for the biostatistician also .
  However, Care Provider cannot be blinded due to the fundamentally different surgical procedures in the three groups. It is not possible to blind the participants since those in the test groups will undergo a specific intervention that involves venous blood withdrawal for the preparation of PRF and ALB-PRF.
  Concerning the blinding of participants, we will implement partial blinding, which will apply exclusively to the test groups (group 1 and 2) involved in a specific intervention that requires venous blood collection for the creation of PRF and ALB-PRF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- empty socket (Other)
  Interventions: Other: empty socket
- Autogenous Dentin Graft with Platelet Rich Fibrin (Active Comparator)
- Autogenous Dentin Graft with Albumin Platelet Rich Fibrin (Experimental)
  Interventions: Procedure: Autogenous Dentin Graft with Albumin Platelet Rich Fibrin

INTERVENTIONS:
Other: empty socket — Patients will be left socket empty without any graft materials for spontaneous healing process after tooth extraction
  Arms: empty socket
Procedure: Autogenous Dentin Graft with Platelet Rich Fibrin — Patients will be inserting autogenous dentin graft and platelet rich fibrin in the socket after extraction.
Procedure: Autogenous Dentin Graft with Albumin Platelet Rich Fibrin — Patients will be inserting autogenous dentin graft and Albumin Platelet Rich Fibrin in the socket after extraction.
  Arms: Autogenous Dentin Graft with Albumin Platelet Rich Fibrin

SUMMARY:
The study focuses on the impact of tooth loss on alveolar bone, which shrinks significantly within the first three months. To prevent this, strategies like alveolar ridge preservation are used.

Autogenous dentin, taken from the patient, supports healing and bone regrowth. Platelet-rich fibrin (PRF), made from the patient's blood, enhances healing and bone density by releasing growth factors.

A new technique combining L-PRF with albumin creates a stable healing membrane that provides a steady release of growth factors. Overall, these methods improve recovery after tooth extractions and prepare sites for future dental work.

DETAILED DESCRIPTION:
Study Design and Randomization:

* Patients classified randomly using computer-generated randomization.
* Performed by the supervisor.
* Three main study groups established.
* Decision for treatment group assignment based on randomized numbers in opaque sealed envelopes, picked by the supervisor.

Groups:

1. Control Group:

   * 20 sockets with empty sockets to allow spontaneous healing post-extraction.
2. Study Group 1:

   * 20 sockets receiving autogenous dentin graft and platelet-rich fibrin (PRF) block.
3. Study Group 2:

   * 20 sockets receiving autogenous dentin graft and Albumin PRF (Alb-PRF) block.

Materials and Preparation

1. Autogenous Dentin Graft:

   The tooth that has been removed will be thoroughly cleaned of any leftover periodontal ligaments, cementum, soft tissue connections, decay, or restorations using a high-speed fine finishing stone along with saline irrigation. Using sterile endodontic files, the pulp chamber will thoroughly be cleaned. Subsequently, the tooth will be ground using a Dentin grinding device to achieve a particle size between 300-1200 μm .The Autogenous Dentin Graft particles will be prepared by demineralizing tooth graft particles through immersion in 0.6N hydrochloric acid for 30 minutes. This will be followed by two rinses with saline and drying with sterile gauze.
2. Platelet-Rich Fibrin (PRF):

   A sample of 10 ml intravenous blood will be collected from the median antecubital vein of the patient. This blood will be placed in 10 ml glass tubes without any additives and will be immediately centrifuged at 3000 RPM for 10 minutes at room temperature. The tube will be separated into three parts, namely, a packed red blood cell at the bottom, acellular plasma at the top, and the PRF clot in between. The PRF clot will be extracted from the tube with the help of sterile tweezers and a surgical blade and then placed in the PRF box to obtain a membrane.
3. Albumin Platelet Rich Fibrin (Alb-PRF):

Nine milliliters of blood in plastic tubes will be centrifuged at 700 g for 8 minutes using an Eppendorf centrifugate. The upper layer (platelet-poor plasma layer) was collected in 2-mL syringes and heated at 75°C for 10 minutes to create denatured albumin (albumin gel). Following heating, the albumin gel was allowed to cool to room temperature for 10 minutes. Then, liquid PRF including remaining cells and growth factor found within the buffy coat layer was thereafter mixed back together with the cooled albumin gel to form Alb-PRF using a female-female luer lock connector. This combination allowed that both the lower-resorption properties of the albumin gel along with the higher cell content and growth factor content of the liquid PRF layer to be remixed. The injectable Alb-PRF gels will then be transferred into culture plate forming a gelated ALB-PRF membrane.

Preoperative Evaluation:

* Clinical examination to confirm eligibility.
* Full mouth charting for periodontal evaluation.
* Patient education on plaque control and oral hygiene.
* Supra & subgingival debridement performed.

Clinical Procedure:

* Pre-extraction rinse with 0.12% chlorhexidine.
* Local anesthesia using 2% mepivacaine HCL with levonordefrin.
* Tooth extraction via minimally traumatic flapless technique.
* Evaluation of extraction socket integrity.

Post-Extraction Treatment

* Control Group: Left the socket empty for healing.
* For the Autogenous Dentin Graft with Platelet Rich Fibrin Block group:

Use surgical curved scissors to cut the two L-PRF membranes into very small pieces, mix chopped membranes and dentin substitute in Ti-dish (2 membranes / 0.5g dentin graft), Add 1 cc of liquid fibrinogen to the homogeneous mixture and gently stir for 5 to 10 seconds while shaping it into the desired form, Fibrinogen will clot into fibrin within a few minutes and trap the biomaterial to form a L-PRF block. the graft will be placed into the socket and will be Covered with a PRF membrane and secured with a single crisscross 5-0 polypropylene suture.

- For the Autogenous Dentin Graft with Albumin Platelet Rich Fibrin group: Mixing the autogenous dentin particles with ALB-PRF in a 1:1 ratio to create a cohesive graft material (dentin block). The graft material is now fully prepared for use. the graft will be placed into the socket and will be Covered with a gelated ALB-PRF membrane. sutured by a single crisscross 5-0 polypropylene suture.

Postsurgical Care Instructions:

1. Avoid Trauma: Do not disturb the surgical site or sutures.
2. Diet: Avoid hot food and refrain from rinsing your mouth.
3. Oral Hygiene: Do not brush the surgical area for 2 weeks; gentle brushing can resume afterward.
4. Medications:

   * Take Amoxicillin 500mg three times daily for 10 days or Doxycycline 100mg twice daily if allergic to penicillin.
   * Use Ibuprofen 600mg for severe pain as needed.
5. Mouthwash: Use a 0.12% chlorhexidine mouthwash for gentle rinsing, twice daily for 2 weeks.
6. Postoperative Issues: Contact your physician immediately if you experience abnormal bleeding.
7. Suture Removal: Sutures will be removed 2 weeks after surgery.
8. Follow-up: Schedule a follow-up appointment 6 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients.
* Adult patients above 18 Years to 60 Years.
* Non-restorable tooth indicated for extraction.
* Posterior mandibular teeth.
* Inactive infection related to the tooth.
* Cooperative patients.

Exclusion Criteria:

* Presence of any systemic disease that could influence the outcome of the therapy.
* Presence of any risk factor (smoker, pregnant and lactating patients).
* Patients with bone diseases.
* Patients with poor oral hygiene.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge width (buccolingual). | at baseline immediately after extraction and after six months
  Will be assessed via Cone-Beam Computed Tomography (CBCT) that Provides a radiographic assessment of the buccolingual width by measuring the distance between buccal and lingual bone walls.
Alveolar ridge height (apicocronal) | at baseline immediately after extraction and after six months
  Will be assessed via Cone-Beam Computed Tomography (CBCT) that Provides a radiographic assessment of the apicocronal height by measuring the ridge height from the top of the alveolar ridge to the upper border of the alveolar canal.
Bone density | at baseline immediately after extraction and after six months
  Will be assessed via Cone-Beam Computed Tomography (CBCT) The measurement helps in assessing the quality of bone directly through Hounsfield units (HU) (between D1 and D5; D1: > 1250 HU, D2: 850 to 1250 HU, D3: 350 to 850 HU, D4: 150 to 350 HU, D5: < 150 HU).

SECONDARY OUTCOMES:
Pain scores | at 24 hours, 3 days, 7 days and 14 days postoperative
  The patients will report their pain score directly through VAS score (between 0 and 10; 0: no pain, 1: minimal pain, 5: moderate pain, and 10: severe pain).
Patient satisfaction | at 24 hours, 3 days, 7 days,14 days postoperative and after six months
  Will use Surveys/Questionnaires to assess patient satisfaction regarding treatment outcomes and experiences. The patients will report their satisfaction score directly through satisfaction score (between 0 and 4; 0: Very satisfied, 1: Satisfied, 2: Neither satisfied nor dissatisfied, 3: Dissatisfied, 4: Very dissatisfied).
Keratinized tissue width | at baseline before extraction and after six months
  Will be assessed through probing techniques before and 6 months after surgical intervention.
  The measurements will be taken at the vertical distance from a line connecting the two neighboring teeth at the CEJs to the free gingival margin (FGM) using a UNC 15 probe (Nordent Manufacturing Inc., IL, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Enas Ahmed Elgendy, PhD, Study Director — Kaferelsheikh University
Locations (1):
- Kaferelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No